CLINICAL TRIAL: NCT04213014
Title: Guys/Girls Opt for Activities for Life Trial
Brief Title: Guys/Girls Opt for Activities for Life Trial (GOAL) to Increase Young Adolescents' Physical Activity and Healthy Eating
Acronym: GOAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lorraine Robbins, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002538; R61HL144896 (NIH); R33HL144896 (NIH)
Record Dates: First submitted 2019-12-20; First posted 2019-12-30 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Adolescent
Keywords: exercise; nutrition; parent; adolescent; overweight; percent body fat; cardiorespiratory fitness; body mass index; obesity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The 16-wk intervention has 3 components.
  1. After-School GOAL Club for moderate-to-vigorous physical activity (MVPA) and healthy eating/cooking skill-building (13 weeks; 120 min/event [N=26]; 2 days/week; not offered for 3 weeks of holiday, winter, spring school breaks).
  2. Three Parent Meetings to empower participants regarding physical activity (PA) and healthy eating and cooking (90 min/meeting [N=3]; Weeks 1, 6, & 11).
  3. GOAL Social Networking Website for Parents to help their adolescents with MVPA and healthy eating and cooking (parents will complete weekly healthy habit-forming tasks; Weeks 1-16). The website will offer information, encouragement, and behavioral strategies to help parents increase their adolescents' PA and healthy eating.
Who Masked: Outcomes Assessor
Masking Description: After baseline data collection, adolescents and parents at each school will be told whether they will receive the GOAL intervention or not. We see no way to blind participants as to which group they are in. Adolescents, parents, principals, school staff, interventionists, and process evaluators will not be told about study aims and hypotheses. Process evaluators (trained by Co-I Pfeiffer) will be independent and not involved in other study areas. Data collectors and biostatistician will not be aware of any adolescent's or parent's (the dyad's) randomization status. Data collectors and interventionists are in separate teams and have separate training and meetings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guys/Girls Opt for Activities for Life Intervention (GOAL) (Experimental): Receives the 4 month (16-wk) GOAL intervention, which has 3 components: (1) After-school GOAL Club: 26 events (2 d/wk; 120 min/event/day; 13 wks due to no club during 3 school break wks) for boys and girls to engage in physical activity and healthy eating and cooking activities; (2) Three parent-adolescent meetings (1st meeting at each school with parents and adolescents [Zoom option if needed]; 2nd and 3rd meetings delivered virtually for parents): to empower parents to assist adolescents with physical activity and healthy eating and cooking; and (3) GOAL social networking website: private website for parents to share with each other how they helped their adolescent increase physical activity and diet quality each week.
  Interventions: Behavioral: Guys/Girls Opt for Activities for Life (GOAL)
- Control (No Intervention): Received usual school activities.

INTERVENTIONS:
Behavioral: Guys/Girls Opt for Activities for Life (GOAL) — The 4 month (16-wk) GOAL intervention has 3 components: (1) After-school GOAL Club: 26 events (2 days/week; 120 min/event/day; 13 weeks due to no club during 3 school break weeks) for boys and girls to engage in physical activity and healthy eating and cooking activities; (2) Three parent-adolescent meetings (1st meeting at each school for parents and adolescents [Zoom option if needed]; 2nd and 3rd meetings delivered virtually and asynchronously for parents): to empower parents to assist adolescents with physical activity and healthy eating and cooking; and (3) GOAL social networking website: private website for parents to share with each other how they helped their adolescent increase physical activity and diet quality each week.
  Arms: Guys/Girls Opt for Activities for Life Intervention (GOAL)

SUMMARY:
In this 2-phase trial (R61/R33), we propose Guys/Girls Opt for Activities for Life (GOAL). Guided by Self-Determination Theory and the Information-Motivation-Behavioral Skills Model, GOAL will target the school and home environment to increase young adolescents' physical activity (PA) and healthy eating by increasing important factors at the individual-level: motivation and self-efficacy; and socioenvironmental-level: social support. The 4-month (16-wk) GOAL intervention has 3 components: (1) After-school GOAL Club: 26 events (2 d/wk; 120 min/event/day; 13 weeks due to no club during 3 school break weeks) for boys and girls to engage in PA and healthy eating/cooking activities; (2) Three parent-adolescent meetings (1st meeting at each school, which is also conducted synchronously via Zoom to increase convenience for parents who are not able to meet in-person at the school for various reasons; 2nd and 3rd meetings video-recorded and delivered asynchronously to accommodate and meet the needs of busy parents who have varying schedules due to work, home, and other responsibilities): to empower parents to assist adolescents with PA and healthy eating/cooking; and (3) GOAL social networking website: private website (already developed) for parents to learn about healthy eating and PA, network with other parents, and share with each other about how they helped their adolescent(s) increase PA and diet quality each week.

The purpose of this individual randomized controlled trial (unit of assignment is adolescent) is to evaluate the effect of GOAL on decreasing cardiovascular disease risk factors (high percent body fat, overweight/obesity, low cardiovascular fitness), improving quality of life; and increasing motivation, self-efficacy, and social support to increase moderate-to-vigorous PA and diet quality among adolescents (5th-8th grade) throughout the state of Michigan. All interested adolescents who meet eligibility criteria and have parental consent will be included. We are including all interested students and not only those who have a high BMI (e.g., BMI z-score ≥0 [≥50th percentile]), in order to avoid social stigma(s) discouraging adolescents from participating. Adolescents in each of 14 schools total will be randomly assigned to the intervention or control (usual school activities) condition. The plan is to include at least n=33 intervention and n=30 control adolescents in each school every year for 3 years of the R33 Phase. On average, we will include at least 63 adolescents per school (at least 31-32 boys and 31-32 girls) and one parent per adolescent will be enrolled, bringing our total sample size to at least 882 dyads total (882 adolescents and one parent per adolescent).

DETAILED DESCRIPTION:
The Guys/Girls Opt for Activities for Life (GOAL) Trial will use an individual randomized controlled trial (IRCT) design. On average, we will include at least 63 adolescents (at least 31-32 boys and 31-32 girls) in each of 14 schools. Adolescents in each school are randomly assigned by our senior biostatistician to either the 16-wk GOAL intervention or a routine school offerings control condition. One parent/guardian (for brevity sake, referred to as parent) per adolescent will also participate as a support person. During each of the 3 intervention yrs (Yrs 3, 4, & 5), the cohort of adolescents and parents participating will differ (Yr 3 Cohort: 4 schools; Yrs 4 & 5 Cohorts: 5 different schools in each year). Data will be collected at 3 time periods from each cohort: 1) pre-intervention/baseline (Wk 0); 2) immediately post-intervention (after 4 months), and 3) 9-month post-intervention follow up (F/U; 13 months post-baseline). We will include, on average, at least 63 adolescents in 5th-8th grade (10-14 yrs old) per school in low-income urban communities in Michigan and one parent per adolescent as a support person. Approximately half of the adolescent participants in each school will be boys, and half will be girls.

R61 Phase (1 year, but extended to 2 years from 2019-2021 due to COVID-19):

Human Subjects approval will be granted from Michigan State University (MSU) Institutional Review Board prior to recruitment. Each school administrator will be asked to identify a program champion to assist researchers during the study.

The PI and Project Manager (PM) will work with the University of Michigan Center for Health Communications Research (CHCR) to make minor refinements to our already developed GOAL social networking website (designed to assist parents in helping their adolescents increase physical activity [PA] and healthy eating) and integrate it into an administrative console with databases for tracking and monitoring day-to-day study operations.

Prior to recruitment, data collection, and the intervention start in fall of Yr 3, the protocol was provided to all permanent research staff for review within the first month of their hire date and prior to any contact with participants.

R33 Phase (Yrs 3-6): R33 was received in 2021; however, study had to be stopped in fall 2021 due to COVID-19 variant and the increased number of positive cases in Michigan that resulted in school closures and restricted access. Individuals external to the schools were not able to enter some schools, and access to students in the schools was limited.

In fall of 2022 (Yr 3), we enrolled 218 adolescents and 1 parent per adolescent who was willing to be a support person from 4 schools. In fall of 2023 (Yr 4), we enrolled 341 adolescents and 1 parent per adolescent who was willing to be a support person from 5 schools. In fall of 2024 (Yr 5), we enrolled 376 adolescents and 1 parent per adolescent who was willing to be a support person from 5 schools. Our biostatistician randomly assigned the adolescents in each school to the intervention or control (usual school activities) condition.

Before the start of school, the research team attended School Open Houses, Orientations, Locker Days, Meet the Teacher Nights, and other events to inform parents and adolescents about the GOAL Project and to distribute a flyer to parents and adolescents about the study. The flyer contained a QR code that linked adolescents to the assent form, parents to the consent form, and both to an eligibility screening tool and baseline survey. At the beginning of each academic school year, the PM, Measurement Coordinator and/or Intervention Coordinator shared study information with 5th-8th grade adolescents at a recruitment assembly at their respective schools. The assembly was hosted in the school for this particular study to invite adolescents to participate. During the assembly, the research team presented the purpose and content of the study and explained details about the after-school program, as well as eligibility requirements for participation. The research team handed out the QR-code-containing flyer to adolescents and asked them to share the information and flyers with their parents. Parents also received an email from each school's administration to share information about the study and invite them to participate with their adolescent. The email included the flyer and QR code so that they could link directly to the assent form, consent form, eligibility screening tool, and baseline survey. Adolescents were told that an adult chosen by the parent would be allowed to serve as the support person if their parent was unable to participate. Parents and adolescents were asked to complete the forms online, if interested in participating, within 4-5 days because registration closed on the 5th day. As schools were initiated in a staggered manner, the research team might also attend a variety of other school events throughout the school year, such as sporting events, parent-teacher conferences, and more. During these events, the research team informed parents and adolescents about the GOAL Project, distributed the QR-code-containing flyer, and invited parents and adolescents to participate in the program.

If acceptable to school administrators, the school's social media site (e.g., Facebook page), email, or text messages were used to inform parents and adolescents about the study and invite them to participate. A link was provided for parents and adolescents to complete forms online. Recruitment also occurred at lunch, during study or library periods, and in classrooms or other venues (depending on permission granted by the school administrators). A 90-second video was been made and shown at the school during assemblies and/or on social media pages. Flyers about the study with a QR code were available in classrooms or other areas in the school for adolescents to take home. The QR code could be used by those interested in participating to easily access study information and complete forms (as noted above). Strategies used might vary in each school depending upon the permission and recommendations received from school administrators.

Response rates were recorded. If far more than enough dyads met eligibility criteria, the PM closed enrollment and capped the number of participating dyads. Although not expected, if an acceptable number of adolescents in a school did not meet eligibility criteria (after several recruitment attempts) or an acceptable number was not reached, the research team recruited higher numbers of participants in subsequent schools. Once enrollment was closed, the study biostatistician randomly assigned the adolescents and parents in each school to the intervention or control (usual school activities) condition. No changes to enrollment or group assignment occurred once randomization was complete. If any participants dropped out before baseline data collection, they were recorded as lost to baseline data collection

Once randomization was completed, the PM contacted all eligible parents to inform them that they and their adolescent were included in the study, based on the eligibility criteria and number of participants needed. Parents were informed that data collection would occur for their adolescents during the school day at baseline, post-intervention, and 13 months post-baseline (9-month F/U). Adolescents completed questionnaires online to assess their perceptions related to PA and healthy eating at baseline and post-intervention. At all 3 time points, quality of life was assessed; and height, weight, % body fat were obtained. At baseline and post-intervention, adolescents' moderate-to-vigorous physical activity (MVPA) via accelerometer was measured, and they completed cardiovascular fitness testing at school. Two 24-hour dietary recalls (1 weekday; 1 weekend day) were conducted with only the adolescents by phone at baseline and post-intervention. To reduce parent burden, stress, and strain (noted by principals due to both the pandemic and inflation), only subjective (self-reported) online survey data were collected from parents. Parents completed an online survey at baseline and post-intervention; and also reported their height and weight at baseline, post-intervention, and 9-month F/U. Therefore, we were not able to measure percent body fat on the parents.

After baseline data were collected, the PM contacted parents to inform them of their group assignment (the GOAL intervention group or GOAL control group). Parents and adolescents in the control condition were told that in a little over 4 months, they would be contacted for data collection and again in the next school year for 9-month F/U. Both groups would receive compensation for participation in data collection.

In November-December of Years 2022 (Yr 3), 2023(Yr 4), and 2024 (Yr 5), the 16-wk intervention began in 4 schools, 5 schools, and 5 schools, respectively, for a total of 14 schools. Parents and adolescents in the intervention group were asked to select 1 of 2 dates and times to attend Dyad Meeting 1 (occurred in Week 1 of intervention; 90-min event) at their adolescents' school (or via Zoom if necessary for those who could not attend in-person) to receive information about the intervention. To accommodate family schedules, the same meeting occurred at 2 time points. During Dyad Meeting 1, the PM and/or Intervention Coordinator presented a study overview. Information, along with behavioral and communication strategies, to assist parents in helping their adolescent increase healthy eating and PA were discussed. A GOAL Club behavioral code of conduct was discussed. Each parent received a GOAL Parent Manual and cookbook. A video of a chef (prepared in R61 Phase) was shown. This video is one of six total (3 for parent-adolescent meetings; 3 for the club) showing the chef conducting a healthy eating and cooking lesson. Finally, parents were assisted with accessing and using the GOAL social networking website. After Dyad Meeting 1, each parent received an Amazon gift card for attending the 1st parent-adolescent meeting.

After Dyad Meeting 1, the 16-week GOAL social networking website intervention component for parents began. It included the 3 weeks during school holiday/winter/spring breaks (every week for 16 weeks). We only included parents with adolescents at the same school in their own private group on the website. To assist parents in increasing their adolescents' PA and healthy eating, we posted an attractive flyer on the website that is focused on a different theme for parents each week, which also aligned with the themes the adolescents were learning in the after-school club. Each theme included: 1) information about PA and healthy eating; 2) 2-3 behavioral strategies related to the information received; and 3) a motivational message. Parents were asked to complete weekly habit-forming tasks regarding how they helped their adolescents with PA and healthy eating/cooking. Each weekly healthy habit-forming task had 3 parts: 1) Parents were asked to post at least one photo or comment about how they helped or planned to help their adolescents with healthy eating/cooking or PA during the week. 2) They were asked to respond to 2 multiple choice questions (one on PA; other on healthy eating) based on the week's flyer information. 3) They were encouraged to respond to at least 1 other parent posting on either PA or healthy eating or cooking with a positive comment.

On Wednesday mornings, parents received information on the upcoming week's healthy habit-forming tasks. Those who did not complete the week's healthy habit-forming task received a text message reminder every day until the task was completed. Once completed, text reminders ceased. If a parent did not complete the weekly tasks consistently, a RA contacted the parent by phone to discuss any barriers preventing the completion of the tasks. Trained RAs monitored site activities, usage, and all postings. RAs responded with a positive comment to all parents who posted about PA and healthy eating. The weekly theme that parents were focusing on was discussed with adolescents at the beginning of the respective healthy eating/cooking and PA sessions offered in the GOAL Club every week. Each week via the website, we posted GOAL Club recipes of the week, information about PA and healthy eating/cooking skills offered in the club, and pictures for parents to see adolescents engaging in club activities if available. The CHCR managed data from the website.

The after-school GOAL Club occurred 2 days/week for 13 weeks (26 120-minute events over the course of 13 weeks; not conducted during school holiday/winter/spring breaks). We employed 5 club instructors/coaches (2 for PA session [1 male; 1 female]; 2 nutrition educators [1 male; 1 female]) and 1 manager [e.g., those who had education and/or experience conducting PA and nutrition programs for adolescents]). We planned to hire and train MSU undergraduate students to serve as coaches for the PA and nutrition program. At least 1 instructor present at each club session was certified in first aid and cardiopulmonary resuscitation. Each adolescent was expected and encouraged to attend the club 2 days every week (total 26 events).

The first 5 min of the 120-min club will included: organizational tasks, healthy snack, and receipt of a motivational message to encourage PA and healthy eating and promote positive perceptions. To increase the comfort level of each group during PA, boys and girls were separated into 2 groups so 1 group could attend the PA session, while the other attended healthy eating and cooking skill-building. Gender non-conforming adolescents were able to choose which group to participate with. Either group began with PA, then switched to the healthy eating/cooking skill-building session and vice versa.

The 50-min "hands on" healthy eating/cooking skill-building session was conducted by 2 nutrition coaches. The session began with a discussion of the healthy eating/cooking weekly theme, as well as information and behavioral strategies that parents were receiving via the GOAL social networking website. Each week during the 1st club day, adolescents were asked to share healthy foods eaten or cooked during the past week when not at the club; on the 2nd day, adolescents were asked to share what they plan to do to eat healthy over the next several days until returning to the club. Adolescents were involved in a healthy eating/cooking skill-building session (45-50 min). Mobile kitchens and our GOAL Club Healthy Eating & Cooking Skill-Building Curriculum was used. Adolescents were able to sample their prepared healthy beverage, snack, or meal.

The 50-min PA session included: 5 min for PA weekly theme discussion, including information and behavioral strategies that parents were receiving via the GOAL social networking website. Each week during the 1st club day, adolescents were asked to share PAs engaged in during the past week when not at the club. On the 2nd day, adolescents were asked to share what they plan to do to attain PA over the next several days until returning to the club. After the discussion, they engaged in 10 min of dynamic warm-ups and fun physically active games; 20 min of sport skill-building; 10 min of fun physically active game(s) to apply learned sports skills; and 5 min of static stretching. Our PA Curriculum was followed as closely as possible, based on available space and resources at the school(s).

In the final 5 minutes of the club, each adolescent was provided with a snack that they could enjoy while completing 4 multiple-choice questions (to evaluate information provided) that served as dose-received data collection. During dismissal, students were compensated $5 for their dose-received data collection. After the club, adolescents were: (1) released to walk home if approved by parents, (2) picked up by parents, or (3) transported home by school bus.

In Week 6 of the intervention (Meeting 2: recorded asynchronous video session), a Co-I reviewed nutrition labels, why they were required, and what information they contained. Nutrition facts on fats, cholesterol, sodium, sugar, and proteins were shared to encourage parents to review the labels when purchasing groceries. Healthy cooking tips, suggestions to select healthy foods at restaurants, and techniques to encourage adolescents to maintain healthy eating were also presented. The chef's video on healthy eating/cooking and preparing a healthy meal was also shown.

In Week 11 (Meeting 3: recorded asynchronous video session), a Co-I reviewed information and behavioral strategies for helping parents continue to assist adolescents in maintaining PA. The session began by discussing how to start the PA journey slowly. SMART goals, good form walking, warming up and stretching were introduced. A video that demonstrated "good form" walking was shown as well. The Co-I presented information on moderate and vigorous physical activity, what the differences are between the two types of PA, and how often adolescents and parents should engage in them per week. Suggestions on how to optimize PA both indoors and outdoors, how to improve sleep and become more physically active overall was provided.

In an intervention conclusion email, the dyads were thanked for their time and effort throughout the GOAL intervention, encouraged to continue their healthy eating and PA behaviors, and provided with a pamphlet containing local community resources, activities, and more.

The intervention ended in 4 schools in early spring 2023 (Yr 3), 5 schools in early spring 2024 (Yr 4), and 5 schools (Yr 5) in early spring 2025 (Yr 5). Post-intervention data collection for parents and adolescents in the schools immediately followed the intervention. In Yr 4, parents and adolescents in the 4 schools of Yr 3's intervention completed the 9-month post-intervention F/U data collection (13 months post-baseline). In Yr 5, parents and adolescents in the 5 schools of Yr 4's intervention completed the 9-month post-intervention F/U data collection (13 months post-baseline).

In Yr 6, parents and adolescents in the 5 schools of Yr 5's intervention will complete the 9-month post-intervention F/U data collection (13 months post-baseline). Procedures will be similar to those used for the schools beginning the study in Yrs 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

Adolescent inclusion criteria are:

1. 5th-8th grade boys and girls (ages 10-14)
2. available and willing to participate in GOAL, including the school club conducted after school 2 days/week for 13 weeks (not during 3 weeks of school breaks)
3. available for follow up (9 months after intervention ends)
4. agree to random assignment
5. able to read, understand, and speak English or have an interpreter
6. able to identify one parent/guardian who is willing and able to serve as a support person and complete study activities

Adolescent exclusion criteria are:

1. mental or physical health condition precluding safe MVPA
2. taking medications that alter appetite, weight, or growth.

Parent/guardian inclusion criteria are:

1. have male or female student in 5th-8th grade
2. ≥18 yrs. of age
3. available and willing to participate in GOAL
4. able to read, understand, and speak English or have an interpreter
5. have Internet access and device for accessing website (e.g., mobile phone ["smart" phone], tablet, computer) and a cellphone which can receive text messages.
6. mentally and physically able to serve as a support person.

Parent/guardian exclusion criteria are:

1. mental or physical health condition precluding engagement in safe MVPA and healthy meal preparation with adolescent
2. not interested in using a private social networking website, similar in design to Facebook, to respond to challenges
3. not interested in learning to post.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — In each school, boys and girls (on average, at least 63 adolescents per school; approximately 1/2 boys and 1/2 girls) and one parent/guardian per adolescent (male or female who is willing to serve as a support person) will be included.
Enrollment: 935 (Actual)
Dates: Start 2020-09-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Percent (%) Body Fat (adolescents) to 4 months (immediate post-intervention) and to 13 months post-baseline (9-month post-intervention follow up [F/U]) | baseline (0 months), immediately post-intervention (after 4 months), and 9-month follow up (13 months post-baseline)
  Bioelectric impedance analysis (BIA) will be used to estimate % body fat. The manufacturer's protocol will be followed (RJL Quantum [IV] BIA Systems, Clinton Township, MI). Testing will be conducted behind a privacy screen by 2 data collectors. Boys and girls will void before testing. Measures will be taken with electrodes: 1 placed on the hand, wrist, foot, and ankle; all on right side of body. Percent (%) body fat will be measured to nearest .1%. Two measurements will be taken. Results are available immediately from the RJL software program. If the 2 measurements differ by >1%, a 3rd measurement must be taken.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) and Overweight/Obesity Percentage from baseline to 4 months (post-intervention) and to 13 months post-baseline (9-month post-intervention follow up [F/U]). | baseline (0 months), immediately post-intervention (after 4 months), and 9-month follow up (13 months post-baseline)
  Two data collectors will measure each adolescent behind privacy screen. Ht without shoes will be measured to nearest 0.10 cm with a stadiometer. Data collectors will position adolescent next to the stadiometer board with head in the Frankfurt horizontal plane. Wt in kg to nearest 0.10 kg will be measured using a foot-to-foot bioelectric impedance scale. Two measurements will be taken for ht and wt. If the 2 differ by <0.5 cm and <0.5 kg, they will be averaged to determine final ht and wt, respectively. If the 2 ht measurements differ by ≥0.5 cm and wt measurements differ by ≥0.5 kg, a 3rd one will be taken. If the 3rd measurement is ≥0.5 cm or ≥0.5 kg. different from the other 2, process will be repeated and another RA will measure. Wt and ht will be combined to estimate BMI for age and sex and overweight/obesity percentage by using the Statistical Analysis System/Software program for Centers for Disease Control and Prevention (CDC) Growth Charts.
Change from Baseline Cardiovascular (CV) Fitness (adolescents) to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  The Progressive Aerobic Cardiovascular Endurance Run (PACER), a 20-meter shuttle run, will be used to estimate aerobic capacity and CV endurance. Guided by a PACER Compact Disc (CD), adolescents will run as long as possible back and forth across a 20-meter or 15-meter (if 20-meters not available) flat surface at a pace that gets faster each min. A lap is one 20-meter or 15-meter distance (from one end to the other). Two RAs will mark the testing area with floor tape. RAs will ask no more than 6 adolescents at a time to run from one line to another until they cannot keep up the pace. One RA will be responsible for no more than 3 boys or girls. The scorer will record the total number of laps completed by each adolescent. Scores will be transferred to a laptop computer. A mile equivalency value will be determined and entered into an equation, according to recommendations. CV fitness is assessed via estimation of maximal oxygen consumption (VO2max).
Change in Minutes of Moderate-to-Vigorous Physical Activity (MVPA; adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  The ActiGraph triaxial (GT3X-plus and wGT3X-BT) accelerometer will record acceleration counts from which min of MVPA will be estimated (analysis software available). Instructions will be provided: right hip (attached to belt) from time getting out of bed in morning to time returning to bed at night for 7 consecutive days. To remind each adolescent to wear it, each will receive a text message (phone call if preferred) at home every morning. Monitors will be initialized and set to begin data collection at 5 o'clock in the morning on the day after they are distributed to adolescents at school. Adolescents will return monitors at school after the 7th day. Data (raw mode, 30Hz) from 7 days will be available for analysis. Data will be downloaded to the same computer used to initialize monitors. To determine intensity, data will be processed using the GGIR package in R with Hildebrand hip-based, ENMO thresholds.
Change in Quality of Life (adolescents) from baseline to 4 months (immediate post-intervention) and to 13 months post-baseline (9-month post-intervention follow up [F/U]). | baseline (0 months), immediately post-intervention (after 4 months), and 9-month follow up (13 months post-baseline)
  The 23-item Pediatric Quality of Life Inventory (Peds QL), which will be used to measure adolescents' health-related quality of life, consists of 4 domains: physical (8 items), emotional (5 items), social (5 items), and school (5 items). Adolescents will respond to a 5-point Likert scale (0 = never; 1 = almost never; 2 = sometimes; 3 = often; 4 = almost always) to indicate how much of a problem each item has been for them during the past month. Items are reverse-scored and transformed to a 0 - 100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) so that the higher the score, the better the quality of life.
Change in Diet Quality (e.g., healthy eating index, servings of fruit and vegetables, sweetened beverage consumption; adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  Adolescents will complete 2 non-consecutive 24-hr dietary recalls (1 weekend day; 1 weekday; randomly selected) over 2-3 weeks at baseline and post-intervention. The Minnesota Nutrition Data System for Research (NDSR) will assess diet quality and obtain a healthy eating index score. Trained staff will collect data from each adolescent via telephone. Adolescents unable to be reached by phone will be contacted at school to complete recalls. To aid in assessing portion sizes, 2-dimensional food models and measuring guides will be given to adolescents at school. The 24-hr recall method, including phone interviews, has been validated in children. The NDSR software will be used to conduct full dietary analysis. Data will be analyzed by the Coordinating Center.
Change in Physical Activity Self-Efficacy (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  A 6-item Perceived Physical Activity Self-Efficacy Scale will be used to assess adolescents' confidence in overcoming barriers (e.g., I can be active in my free time on most days even when I am busy). Response choices range from: (0) not at all sure to (3) very sure. A higher score means a better outcome.
Change in Social Support for Physical Activity (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  A 8-item Family and 3-item Friend Support Scale will be used to determine adolescents' perceptions of the total instrumental assistance and emotional encouragement for physical activity received from significant others. Response choices range from: (0) never to (5) very often. A higher score means a better outcome.
Change in Motivation for Physical Activity (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  Twelve items from the Behavioural Regulation in Exercise Questionnaire (BREQ-3) will be used to assess adolescents' motivation for PA. Response choices range from: (0) not true for me to (4) very true for me. A higher score means a better outcome.
Change in Self-Efficacy for Healthy Eating (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  A 9-item Child Dietary Self-Efficacy Scale will be used to determine adolescents' confidence related to healthy eating. Response choices are: (0) not at all sure, (1) not very sure, (2) somewhat sure, and (3) very sure. A higher score means a better outcome.
Change in Baseline Social Support for Healthy Eating (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  An 8-item Family (4 items) and Friend (4 items) Support for Healthy Eating Scale will be used to assess adolescents' perceptions of family and friend instrumental assistance and emotional support for healthy eating. Response choices include: (0) never, (1) rarely, (2) sometimes, (3) often, and (4) very often. A higher score means a better outcome.
Change in Motivation for Healthy Eating (adolescents) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  Motivation for healthy eating will be assessed with 12 items from the Regulation of Eating Behaviors Scale. Response choices range from not true for me (0) to very true for me (4).
Change in Family Nutrition and Physical Activity (exploratory aim; parents/guardians) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  Parents/guardians will complete a 20-item Family Nutrition and Physical Activity Screening Tool that will be used to evaluate health behaviors in the home. Response choices range from: (1) never/almost never to (4) very often/always. A higher score means a better outcome.
Change in Minutes of Moderate-to-Vigorous Physical Activity (MVPA; exploratory aim; parents/guardians) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  All parents will complete the International PA Questionnaire. The questionnaire is a 7-day recall of PA behavior. It is used with adults to determine the frequency (days/week) and duration (mins/day) of various activities, such as walking, moderate PA (carrying light loads, bicycling at a regular pace), and vigorous PA (heavy lifting, aerobics, or fast bicycling). Responses will be converted to metabolic equivalent task minutes per week (MET-min/week). Parents will be classified as participating in low, moderate, or high levels of PA based on a scoring protocol.
Change in Diet Quality (exploratory aim; parents/guardians) from baseline to 4 months (immediate post-intervention) | baseline (0 months) and immediately post-intervention (after 4 months)
  All parents will complete the 10-item Block Fruit-Vegetable-Fiber Screener. Responses range from: (1) Less than 1/WEEK to (5) 2+ a DAY. A higher score means a better outcome.
Change in Body Mass Index (BMI; exploratory aim; parents/guardians) from baseline to 4 months (immediate post-intervention) and to 13 months post-baseline (9-month post-intervention follow up [F/U]) | baseline (0 months), immediately post-intervention (after 4 months), and 9-month follow up (13 months post-baseline)
  BMI will be calculated based on weight (kilograms)/height (meters squared). Parents/guardians will self-report height and weight for the analysis of BMI.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Data and study documentation materials will be released to the NHLBI and within the timelines described in the NHLBI Policy for Data Sharing from Clinical Trials and Epidemiological Studies. The data sets will be submitted to the study NHLBI Program Official no later than 3 years after the end of the final follow-up or 2 years after the main paper of the trial has been published, whichever comes first.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data sets will be submitted to the study NHLBI Program Official no later than 3 years after the end of the final follow-up or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: We plan to adhere to the NHLBI Policy for Data Sharing from Clinical Trials and Epidemiological Studies and Guidelines for NHLBI Data Set Preparation. Documentation for data sets will be clear to enable other researchers not familiar with a data set to use it in the future. A summary documentation file will be created to provide a complete overview of the data and description of their use for researchers who are not familiar with the data set. Data will only be made available under terms consistent with the informed consent provided by individual participants, and as approved by the Michigan State University (MSU) Human Research Protection Program/Institutional Review Board (IRB) and any local, state, and federal laws and regulations. In addition, de-identified electronic data will be archived in the MSU College of Nursing (CON) for use by faculty, students, or other researchers in the future. Interested users will be asked to contact the PI and sign a data sharing agreement.

REFERENCES:
- [Background] Robbins LB, Ling J, Pfeiffer KA, Kerver JM, Resnicow K, McCaffery H, Hilliard A, Hobbs L, Donald S, Kaciroti N. Intervention to increase physical activity and healthy eating among under-represented adolescents: GOAL trial protocol. BMJ Open. 2024 Jan 3;14(1):e080437. doi: 10.1136/bmjopen-2023-080437. PMID 38171630
- [Derived] Fraczek N, Robbins LB, Varpaei HA, Arcoleo K, Ling J. Relationships of motivation, self-efficacy and social support with healthy eating behaviours among adolescents. BMJ Nutr Prev Health. 2025 Nov 28;8(2):e001369. doi: 10.1136/bmjnph-2025-001369. eCollection 2025. PMID 41502578